CLINICAL TRIAL: NCT04339478
Title: Does Parathyroid Autofluorescence Reduces Unintensional Parathyroidectomy During Total Thyroidectomy with Central Lymph Node Compartment Dissection
Acronym: FLUOBCC
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Umraniye Education and Research Hospital (Other Government); The Hashemite University (Other)
Responsible Party: Principal Investigator, Papavramidis Theodossis, Assistant Professor of Surgery, Aristotle University Of Thessaloniki
Other Study IDs: FLUOBCC
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2021-08

CONDITIONS: Thyroid Cancer; Thyroidectomy with Central Lymph Node Dissection
Keywords: Thyroidectomy; Central Lymph node compartment dissection; autofluorescence; FLUOBEAM XS
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Autofluorescence: The surgeon will perform the preplanned thyroidectomy with central lymph node compartment dissection with FLUOBEAM XS. The following intraoperative variables will be recorded for all patients:
  Surgery date Duration of surgery Operation performed Procedure related comments Number and location of the visualized glands Intra-operative autofluorescence score (either 0 (no visualization or 1 visualization) for each gland
- Control: The surgeon will perform the preplanned thyroidectomy with central lymph node compartment dissection without autofluorescence device. The following intraoperative variables will be recorded for all patients:
  Surgery date Duration of surgery Operation performed Procedure related comments Number and location of the visualized glands

SUMMARY:
The aim of the study is to evaluate the effectiveness of autofluorescence in the intraoperative preservation of parathyroids during total thyroidectomy with central lymph node compartment dissection.

DETAILED DESCRIPTION:
Real-time intraoperative identification and functional maintenance of structures are of major importance in endocrine surgery, with a critical role in clinical outcomes and patients' quality of life. Despite the advances in preoperative imaging techniques, there is still need for precise intraoperative visualizing [1]. Limitations of naked eye inspection and subjectivity of palpation are imposing challenges even for the most experienced surgeons [1-3]. Nowadays, attention is attracted to intraoperative imaging techniques using Near Infrared Fluorescence (NIRF) with endogenous or exogenous contrast agents. These imaging techniques are attractive in biomedicine due to its high penetration depth and low scattering in human tissue [2].

Autofluorescence is the ability of several natural substances or drugs to be fluorescent after the absorbance of light or radiation. It has been already proved that parathyroid glands emit their own light after near-infrared (NIR) around 820nm , providing high contrast to the surrounding tissues. This made near-infrared autofluorescence a potential useful tool in hands of experienced endocrine surgeons in order to distinguish parathyroid glands from other anatomic structures during thyroidectomies.

Approximately 7.6% of thyroid surgeries resulted in hypoparathyroidism, with 75% of these cases being transient and 25% being chronic. The mechanisms that underlie hypoPTH are related to disruption of parathyroid arterial supply or venous drainage, mechanical injury, thermal or electrical injury, and either intentional or inadvertent partial or complete removal.

The aim of the present study is to evaluate the value of intra-operative autofluorescence imaging concerning the unintentional excision rate of parathyroids during total thyroidectomy with central lymph node compartment dissection. Moreover, we are going to evaluate correlation of autofluorescence with 24 hours post-operative PTH.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is over 18 years old
2. Patient scheduled for a non-emergency operation
3. Patient eligible for total thyroidectomy

Exclusion Criteria:

1. Patient is participating in another clinical trial which may affect this study's outcomes
2. Prior operation in the neck
3. Primary or secondary hyperparathyroidism
4. Vitamin D deficiency
5. Use of drugs that influences calcium metabolism (Vitamin D analogues, oral calcium supplements, bisphosphonates, teriparatide, thiazide diuretics, aromatase inhibitors)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Our sample size of 180 patients has been calculated after power analysis regarding other similar studies with an a=0.05 and Power=0.95.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
The contribution of intra-operative autofluorescence imaging on unintentional excision rate of parathyroids during total thyroidectomy with central lymph node dissection | 6 months
  The aim of the study is to evaluate the use of autofluorescence to distinguish parathyroid glands during thyroidectomy with central lymph node dissection (TTCC). We will measure the number of parathyroids accidentally excised during TTCC with and without autofluorescence.

SECONDARY OUTCOMES:
Detecting the changes of practice in performing total thyroidectomywith central lymph node dissection when monitoring parathyroids with autofluorescence. | 6 months
  If autofluorescence is proved to be a useful tool in endocrine surgeons hands, the preservation of parathyroid glands during thyroidectomy with central lymph node dissection would be easier.
Correlating autofluorescence with 24 hours post-operative PTH. | 6 months
  To identify any correlation between intra-operative parathyroid glands autofluorescence with postoperative hypoparathyroidism. We are going to evaluate the number of parathyroids evaluated and we are going to correlate it with PTH.
Correlating autofluorescence with postoperative hypocalcemia | 7months
  To identify any correlation between intra-operative parathyroid glands autofluorescence with postoperative hypoparathyroidism. We are going to evaluate the number of parathyroids evaluated and we are going to correlate it with Ca.
Identifying and analyzing problematic groups of patients | 7 months
  This study will sign out the disadvantages of FLUOBEAM XS or cases that its use should be avoided.

CONTACTS AND LOCATIONS:
Overall Officials: Theodossis Papavramidis, MD, PhD, Principal Investigator — AHEPA University Hospital of Thessaloniki, Greece
Locations (3):
- 1st Propedeutic Department of Surgery, AHEPA University General Hospital, Aristotle University of Thessaloniki, Thessaloniki, Greece
- Department of Surgery, Faculty of Medicine, Hashemite University, Zarqa, Jordan
- Umraniye Education and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No